CLINICAL TRIAL: NCT06749652
Title: Soft Vs. Firm Ureteral Stents: Symptoms Improvement Without Affecting Outcomes- a Prospective, Randomized Trial
Brief Title: Prospective, Randomized Trial Comparing Soft and Firm Ureteral Stents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Orel Hemo, Urology Resident, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0119-23-SMC
Record Dates: First submitted 2024-12-15; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Urolithiasis
Keywords: Urolithiasis; stent-symptoms
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Intervention Model Description: Parallel model has been used. The randomization allocation sequence (1:1) has been generated using asymptomatic maximal randomization. Patients, data collectors and data analysts were blinded to the allocation. As blinding the surgeons during procedure was not possible, they were not involved in either data collection or analysis.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Soft silicone stent arm (Experimental): Patients who recieved soft silicone ureteral stent (Universa, Cook medical) at the end of the ureteroscopy
  Interventions: Device: Soft silicone ureteral stent insertion
- Firm silicone stent arm (Experimental): Patients who recieved firm silicone ureteral stent (percuflex plux, boston scientificl) at the end of the ureteroscopy
  Interventions: Device: firm silicone stent insertion

INTERVENTIONS:
Device: firm silicone stent insertion — Insertion of firm silicon ureteral stent (Percuflex Plus)
  Other Names: percuflex plus
  Arms: Firm silicone stent arm
Device: Soft silicone ureteral stent insertion — Soft silicone ureteral stent insertion
  Other Names: Universa
  Arms: Soft silicone stent arm

SUMMARY:
The goal of this clinical trial is to evaluate whether ureteral stent type impacts stent-related symptoms and quality of life in patients undergoing ureteroscopy (URS) and stone lithotripsy for ureteral stones. The main questions it aims to answer are:

* Does a soft polymer stent reduce stent-related symptoms compared to a firm polymer stent?
* Does stent type affect intra- and postoperative complications? Researchers will compare patients receiving a soft polymer stent (Universa®, Cook Medical) to those receiving a firm polymer stent (Percuflex®, Boston Scientific) to determine if soft stents improve patient comfort and quality of life while maintaining a similar safety profile.

Participants will:

* Undergo URS and stone lithotripsy for ureteral stones.
* Be randomly assigned to receive either a soft or firm ureteral stent.
* Complete the Ureteral Stent Symptoms Questionnaire (USSQ) upon stent removal, 14 days after URS.

DETAILED DESCRIPTION:
Study Design and Patient Selection

1. Study Period and Ethical Approval:

   * Conducted between July 2023 and July 2024 following institutional review board approval (SMC 0119-23).
   * Informed consent obtained from all participants.
   * Adhered to the Declaration of Helsinki.
2. Stent Types and Randomization:

   * Soft stent: Universa® (Cook Medical).
   * Firm stent: Percuflex™ Plus (Boston Scientific).
   * Randomization in a 1:1 ratio using asymptomatic maximal randomization.

Surgical Technique and Intervention Operative Team included three fellowship-trained endourologists.

Procedure Details:

* Ureteroscopy performed using standard 6.5/8.5Fr semi-rigid ureteroscope.
* Lithotripsy performed using a 120W Holmium:YAG laser (0.3 Joule, 40 Hertz, dusting technique).

Stent Placement was performed using a 0.038 Inch glide wire. 6Fr stents used, either soft or firm polymer material, according to randomization.

Proximal stent curls positioned in the upper calyx/renal pelvis; distal curls in the bladder.

Postoperative Care Stent removal was scheduled 2 weeks post-procedure, ans performed using a flexible cystoscope in the outpatient clinic.

Symptoms assesed using the Ureteral Stent Symptoms Questionnaire (USSQ) that was completed at the stent removal visit.

Statistical Analysis

1. Sample Size Calculation:

   * Based on a 3-point difference in USSQ index score between groups.
   * Assumed 5% type I error and 80% power.
   * Adjusted for a 10% dropout rate; target sample size: 140 patients.
2. Data Blinding:

   * Patients, data collectors, and analysts blinded to allocation.
   * Since blinding the surgeons to stent type was impossible, surgeons were not involved in data collection or analysis.
3. Analysis Methods:

   * Continuous variables: Mann-Whitney U test; median and IQR.
   * Categorical variables: Pearson's chi-square or Fisher's exact test; frequencies and proportions.
   * Multivariate linear regression for USSQ index and urinary domain scores.
   * Statistical significance set at p<0.05.
   * Analyses conducted using IBM SPSS v26.

This protocol ensures a rigorous and reproducible methodology for evaluating the impact of stent type on patient-reported outcomes following ureteroscopy and lithotripsy.

ELIGIBILITY:
Inclusion Criteria:

* patients aged over 18 years
* ureteral stones measuring up to 2cm requiring URS and laser lithotripsy

Exclusion Criteria:

* pediatric patients
* bilateral stones requiring bilateral URS and laser lithotripsy,
* stone located in the renal pelvis or calyces,
* intra-operative complications of any kind,
* any residual stones during the procedure,
* ureteroscopies in which no stones were treated ("white ureteroscopy").

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-07-09 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
the Ureteral stent symptoms questionnaire (USSQ )index score | 14 days after stent insertion
  The summation of the Ureteral stent symptoms questionnaire (USSQ) individual question scores. The questionnaire includes 32 questions, with a scale of zero to five points each. The USSQ Index score represents the summation of each indivisual question score, with a scale of 0-160, with higher score means the patients is suffering from more severe symptoms.

SECONDARY OUTCOMES:
Ureteral stent symptoms questionnaire (USSQ) urinary domain score | 14 days after stent insertion
  There are total of 5 different domains in the Ureteral stent symptoms questionnaire (USSQ): urinary synptoms, pain, general health, occupational and sexual distress. The summation of the score of each domain represents a secondary outcome. The urinary domain has 10 questions, each in a scale of zero to five, to a total of 0-50. Higher score means the patient experience more severe urinary symptoms.
Ureteral stent symptoms questionnaire (USSQ) pain domain score | 14 days after stent insertion
  There are total of 5 different domains in the Ureteral stent symptoms questionnaire (USSQ): urinary synptoms, pain, general health, occupational and sexual distress. The summation of the score of each domain represents a secondary outcome. The pain domain has 7 questions, each in a scale of zero to five, to a total of 0-35. Higher score means the patient experience more severe pain.
Ureteral stent symptoms questionnaire (USSQ) general health domain score | 14 days after stent insertion
  There are total of 5 different domains in the Ureteral stent symptoms questionnaire (USSQ): urinary synptoms, pain, general health, occupational and sexual distress. The summation of the score of each domain represents a secondary outcome. The general health domain has 6 questions, each in a scale of zero to five, to a total of 0-30. Higher score means the stent affecting the patients general health in a more prominent way.
Ureteral stent symptoms questionnaire (USSQ) work performance domain score | 14 days after stent insertion
  There are total of 5 different domains in the Ureteral stent symptoms questionnaire (USSQ): urinary synptoms, pain, general health, occupational and sexual distress. The summation of the score of each domain represents a secondary outcome. The work performance domain has 6 questions, each in a scale of zero to five, to a total of 0-30. Higher score means the stent affecting the patients work performance in a more prominent way.
Ureteral stent symptoms questionnaire (USSQ) sexual performance domain score | 14 days after stent insertion
  There are total of 5 different domains in the Ureteral stent symptoms questionnaire (USSQ): urinary synptoms, pain, general health, occupational and sexual distress. The summation of the score of each domain represents a secondary outcome. The sexual performance domain has three questions, each in a scale of zero to five, to a total of 0-15. Higher score means the stent affecting the patients sexual performance in a more prominent way.

OTHER OUTCOMES:
Intraoperative lenght | Upon data collection, at the day of the surgery
  Surgery lenght from the introduction of the ureteroscope to the completion of the stent placment. Measured in minutes.
Postoperative complications | 30 days post discharge
  Postoperative complications reported according to the Clavien-Dindo classification), from the end of the surgery and until 30 days post discharge
Hospitalization length | From hospitalization day until discharge days, collected upon patients' discharge, on average of 1 day
  The total amount of days the patient was hospitalized after the procedure. measured in days.
Emergency department visits | From discharge day to 30 days post discharge
  Total number of emergency department (ED) visits for each patient, wheter they were hospitalized or discharged following that visit.
Number of Re-hospitalizations | From surgery discharge day to 30 days post discharge
  Total amount of re-hopitalization number after the original discharge after the surgery, and until 30 days post discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Kleinmann, M.D., Study Director — Sheba Medical Center, Tel-Hashomer
Locations (1):
- Sheba Medical Center, Ramat Gan, Central District, Israel

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, an anonimized version will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Information will be available after the study will be published, for 2 years
Access Criteria: Upon request to the primary investigator, an anonimized excel sheath will be sent